CLINICAL TRIAL: NCT00697866
Title: Evaluating the Consistency of 3 Consecutive Lots of GSK Biologicals' Novel Adjuvanted HBV Vaccine With Single-blind Safety Evaluation Using Engerix™-B as a Control, Administered According to a 0, 1, 2-month Schedule in Healthy Volunteers (15-50y).
Brief Title: Consistency of 3 Consecutive Lots of a Novel HBV Vaccine With Single-blind Safety Evaluation Using Engerix™-B as Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 208129/037
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Adjuvanted hepatitis B vaccine; Hepatitis B; Recombinant hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): HBV-MPL Lot A
  Interventions: Biological: HBV-MPL vaccine 208129
- Group B (Experimental): HBV-MPL Lot B
  Interventions: Biological: HBV-MPL vaccine 208129
- Group C (Experimental): HBV-MPL Lot C
  Interventions: Biological: HBV-MPL vaccine 208129
- Group D (Active Comparator): Engerix™-B
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — 3 consecutive lots; 3-dose intramuscular injection
  Arms: Group A; Group B; Group C
Biological: Engerix™-B — 3-dose intramuscular injection
  Other Names: HBV-MPL vaccine 208129
  Arms: Group D

SUMMARY:
The purpose of the present study is to evaluate the immunogenicity and safety of three consecutive production lots of the novel adjuvanted HBV vaccine. The safety of the candidate vaccine will be assessed using Engerix™-B as control.

DETAILED DESCRIPTION:
Double-blind for the identity of the consistency lots, single-blind for the control group/study vaccine identity.

At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 15 and 50 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject/ from the parents or guardians of the subject where applicable
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/Administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s).
* Previous vaccination against hepatitis B
* History of non-response to previous hepatitis B vaccination
* Known exposure to hepatitis B within the previous 6 weeks
* History of hepatitis B infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* Suspected or confirmed multiple sclerosis in the subject (applicable to Centre 5/France only)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 951 (Actual)
Dates: Start 2000-08; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody concentrations | At month 3

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | At M1, M2, M3
Anti-RF1 antibody titres in a subset of 50 subjects per group | At months 0 and 3
Occurrence, intensity and relationship to vaccination of solicited local and general signs and symptoms | During a 4-day follow-up after vaccination
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | Within 30 days after each vaccination
Occurrence, intensity and relationship to vaccination of serious adverse events | During the study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 208129/037 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208129/037 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208129/037 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208129/037 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208129/037 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208129/037 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register